CLINICAL TRIAL: NCT03090737
Title: An Open-label, Single-arm Phase II Safety Study of Nivolumab in Participants With Advanced or Metastatic Non-small Cell Lung Cancer Who Have Progressed During or After Receiving at Least One Prior Systemic Regimen (CheckMate 907: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 907)
Brief Title: Safety Study of Nivolumab to Treat Advanced or Metastatic Non-small Cell Lung Cancer
Acronym: CheckMate 907
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-907; 2016-003731-37 (EudraCT Number)
Record Dates: First submitted 2017-03-20; First posted 2017-03-27 (Actual); Results first posted 2022-03-14 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Specified Dose on Specified Days
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Specified Dose on Specified Days
  Other Names: BMS-936558; Opdivo

SUMMARY:
A study to evaluate the safety of Nivolumab in participants with advanced or metastatic non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Non small cell lung cancer (Squamous or non-squamous)
* At least one prior anti-cancer therapy that did not work
* ECOG Performance Scale 0-1

Exclusion Criteria:

* Cancer that has spread to the brain or leptomeninges unless there is no evidence of progression by MRI for 8 weeks after treatment is complete and within 28 days before first dose of study drug
* Active, known or suspected autoimmune disease or infection
* Prior immuno-oncology therapy
* Corticosteroids within 2 weeks of study drug administration

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (5):
  - Alabama Oncology, Birmingham, Alabama
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - St Vincent Frontier Cancer Center, Billings, Montana
  - Broome Oncology, Johnson City, New York
  - Guthrie Medical Group Sayre, Sayre, Pennsylvania
- Canada (3):
  - Local Institution - 0015, Kingston, Ontario
  - Local Institution - 0014, Oshawa, Ontario
  - Local Institution - 0001, Toronto, Ontario
- Japan (4):
  - Local Institution - 0017, Nagoya, Aichi-ken
  - Local Institution - 0023, Osaka, Osaka
  - Local Institution - 0018, Koto-ku, Tokyo
  - Local Institution - 0016, Tokyo
- Romania (2):
  - Local Institution - 0003, Craiova
  - Local Institution - 0006, Sector 2
- South Africa (3):
  - Local Institution - 0011, Port Elizabeth, Eastern Cape
  - Local Institution - 0013, Parktown, Johannesburg, Gauteng
  - Local Institution - 0012, George, Western Cape

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/safety/medwatch/safetyinformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab 480mg Q4W: 480 mg of Nivolumab every 4 weeks (Q4W) until progression, unacceptable toxicity, withdrawal of consent, death, or a max of 2 years, whichever occurs first
Period: Overall Study
Arm/Group | Nivolumab 480mg Q4W
Started (Started=Treated) | 129
Completed | 0
Not Completed | 129
Not completed — Other reasons | 1
Not completed — Completed treatment as per protocol | 17
Not completed — Maximum clinical benefit | 2
Not completed — Adverse event unrelated to study drug | 7
Not completed — Study drug toxicity | 4
Not completed — Disease progression | 98

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab 480mg Q4W
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 26
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 95
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing High Grade (Grades 3-4 and Grade 5) Drug-Related Select Adverse Events (AE)
Description: The number of participants who experienced at least 1 select AE of Grade 3-5, judged to be related to study drug per investigator with onset on or after first dose of study treatment and within 30 days of last dose of study treatment, divided by number of treated participants. AE grade is defined using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0 criteria. The select AEs consist of pulmonary events, gastrointestinal events, hepatic events, renal events, skin events, endocrine events categories, thyroid disorders, diabetes, pituitary, adrenal disorder subcategories. Grade 3 is defined as severe or medically significant but not immediately life-threatening. Grade 4 is defined as life-threatening consequences and urgent intervention indicated. Grade 5 is defined as death related to AE.
Time Frame: From the first dose of study treatment to up to 30 days of the last dose of study treatment (up to 24 months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab 480mg Q4W
Number analyzed (Participants) | 129
Participants
  Total Participants with Grade 3-4 AE | 3
  Total Participants with Grade 5 AE | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time between the date of randomization and the date of the first documented tumor progression accounting for subsequent therapy, based on BICR (blinded independent central review) assessments (per RECIST v1.1 criteria), or death due to any cause, whichever occurs first. Participants will be censored at the last evaluable tumor assessment on or prior to the date of subsequent therapy. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From first dose to the date of the first documented tumor progression (up to approximately 5 months)
Population: All Treated Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 480mg Q4W
Number analyzed (Participants) | 129
Months | 3.68 [3.06 to 4.50]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) defined as the percentage of participants with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) as assessed by investigator per RECIST 1.1. Complete response is defined as the disappearance of all target lesions and the reduction of any pathological lymph nodes to <10 mm. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions. Radiographic tumor assessments will be conducted at Week 8 (+/- 7 days) and every 8 weeks (+/- 7 days) until up to 2 years or until disease progression (or until discontinuation of study therapy in patients receiving nivolumab beyond progression), lost to follow-up, or withdrawal of study consent.
Time Frame: From the date of first dose to the date of the initial objectively documented tumor progression or the date of subsequent therapy, whichever occurs first (up to approximately 25 months).
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab 480mg Q4W
Number analyzed (Participants) | 129
Percentage of participants | 17.1 [11.0 to 24.7]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time between the first dosing date and the date of death due to any cause. For participants without documentation of death, OS will be censored on the last date the participant was known to be alive.
Time Frame: From first dosing date and the date of death due to any cause (up to approximately 4 years and 9 months)
Population: All Treated Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 480mg Q4W
Number analyzed (Participants) | 129
Months | 10.58 [8.34 to 14.69]

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response (DOR) is defined as the time between the date of first confirmed response up to the date of the first documented tumor progression (per RECIST 1.1) as determined by complete response (CR) or partial response (PR), or death due to any cause, whichever occurs first. Participants who neither progress nor die will be censored on the date of their last evaluable tumor assessment. Participants who started any subsequent anti-cancer therapy (including palliative local therapy) without a prior reported progression will be censored at the last evaluable tumor assessment prior to or on the date of initiation of the subsequent anti-cancer therapy (including palliative local therapy). Complete response is defined as the disappearance of all target lesions and the reduction of any pathological lymph nodes to <10 mm. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: From the date of first confirmed response up to the date of the first documented tumor progression (per RECIST 1.1), or death due to any cause, whichever occurs first (up to approximately 48 months).
Population: All Responder Participants (participants with confirmed CR or PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 480mg Q4W
Number analyzed (Participants) | 22
Months | 35.45 [10.87 to 47.31]

6. Post Hoc Outcome: The Number of Participants Experiencing High Grade (Grades 3-4 and Grade 5) Drug-Related Select Adverse Events (AE) - Extended Collection
Description: The number of participants who experienced at least 1 select AE of Grade 3-5, judged to be related to study drug per investigator with onset on or after first dose of study treatment and within 30 days of last dose of study treatment, divided by number of treated participants. AE grade is defined using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0 criteria. The select AEs consist of pulmonary events, gastrointestinal events, hepatic events, renal events, skin events, endocrine events categories, thyroid disorders, diabetes, pituitary, adrenal disorder subcategories. Grade 3 is defined as severe or medically significant but not immediately life-threatening. Grade 4 is defined as life-threatening consequences and urgent intervention indicated. Grade 5 is defined as death related to AE. Note: This outcome measure represents an update to the primary endpoint to include additional data collection that occurred after the primary completion date.
Time Frame: From the first dose of study treatment to up to 30 days of the last dose of study treatment (up to 25 months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab 480mg Q4W
Number analyzed (Participants) | 129
Participants
  Total Participants with Grade 3-4 AE | 6
  Total Participants with Grade 5 AE | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their enrollment to study completion, (up to approximately 4 years and 9 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 27 months)
Arm/Group | Nivolumab 480mg Q4W
All-Cause Mortality (participants affected / at risk) | 105/129
Serious Adverse Events (participants affected / at risk) | 56/129
Other Adverse Events (participants affected / at risk) | 111/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 480mg Q4W (N=129)
Anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Diverticulitis (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pneumonia aspiration (Infections and infestations) | 1
Pneumonia klebsiella (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Influenza A virus test positive (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 37
Amnesia (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 480mg Q4W (N=129)
Anaemia (Blood and lymphatic system disorders) | 37
Hyperthyroidism (Endocrine disorders) | 7
Hypothyroidism (Endocrine disorders) | 8
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 24
Nausea (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 8
Fatigue (General disorders) | 19
Non-cardiac chest pain (General disorders) | 10
Oedema peripheral (General disorders) | 8
Pneumonia (Infections and infestations) | 13
Upper respiratory tract infection (Infections and infestations) | 7
Alanine aminotransferase increased (Investigations) | 12
Aspartate aminotransferase increased (Investigations) | 11
Blood alkaline phosphatase increased (Investigations) | 32
Blood creatinine increased (Investigations) | 11
Weight decreased (Investigations) | 14
Decreased appetite (Metabolism and nutrition disorders) | 21
Hyperglycaemia (Metabolism and nutrition disorders) | 13
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 17
Anxiety (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23
Dry skin (Skin and subcutaneous tissue disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 24
Rash (Skin and subcutaneous tissue disorders) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT03090737/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT03090737/SAP_001.pdf